CLINICAL TRIAL: NCT03382236
Title: Evaluating the Effectiveness of Osteopathy in the Management of Pain in Elderly People in Residential Care Facilities for the Elderly (EHPAD)
Brief Title: Evaluating the Effectiveness of Osteopathy in the Management of Pain in Elderly People
Acronym: IPODE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Léa Gouaux (Other)
Collaborators: BTP RMS (Unknown); ESO Paris Recherche (Other)
Responsible Party: Sponsor-Investigator, Léa Gouaux, Attachée de recherche clinique, Ecole Supérieur d'Ostéopathie
Organization: Ecole Supérieur d'Ostéopathie (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTP RMS
Record Dates: First submitted 2017-12-11; First posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Osteopathy
MeSH Terms: interventions — Osteopathic Physicians

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real osteopathy (Experimental)
  Interventions: Other: osteopathy
- Sham osteopathy (Placebo Comparator)
  Interventions: Other: osteopathy

INTERVENTIONS:
Other: osteopathy — osteopathic techniques

SUMMARY:
This type of study can have an impact on public health policy and help improve the management of pain in people with EHPAD; Propose better use of drug treatments and non-pharmacological methods such as osteopathy; Help structuring the healthcare sector.

DETAILED DESCRIPTION:
* "Osteopathy" group: 3 osteopathy sessions of 45 min with one session every 3 weeks at S2, S5 and S8. Fascial osteopathic techniques performed will consist of gentle and non-impulsive manipulation
* "Simulated" group: 3 simulated osteopathy sessions lasting 45 minutes, one session every 3 weeks at S2, S5 and S8. The techniques performed will consist of an application of the hands to different anatomical regions than the group "osteopathy" without therapeutic intention, that is to say without tissue tensioning.

The pain will be assessed at inclusion (S0) and at the end of the procedure (S12) by the head physician, the coordinating physician or the psychomotor therapist, ignoring the assignment group of the subject and before each session. osteopathy (at S2, S5 and S8) by a nurse or psychomotor also ignoring the patient's assignment group.

Both groups will continue to benefit from their usual allopathic management and recommendations.

Patients will not be aware of the treatment received (osteopathy or simulated) and will be randomized by a computer server.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 75 years
* Patients Residing in Accommodation Facilities for Dependent Old People
* A score measured by the DOLOPLUS 2 Scale at least 7/30 at the start of the study
* For patients in capacity and autonomous: Patients informed and having signed a free and informed consent.

For non-capable patients with a trusted person and / or guardian: Informed patients whose confidant or guardian has been informed and has signed free and informed consent.

- Affiliated to a social security scheme (beneficiary or beneficiary)

Exclusion Criteria:

* Absence of pain
* Medical contraindication known to the practice of osteopathy with fascial aim (advanced degenerative bone disease, metastatic cancer)
* Osteopathic treatment in the last six months
* Patients under curators

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-01-03 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
DOLOPLUS 2 score | Every week after inclusion during 4 weeks
  Assessment of pain assessed by the behavioral scale

CONTACTS AND LOCATIONS:
Locations (1):
- Lea Gouaux, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided